CLINICAL TRIAL: NCT01948063
Title: Ubiquinol (Reduced COQ10) for Patients With Sepsis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Kaneka Medical America LLC (Industry)
Responsible Party: Principal Investigator, Michael Donnino, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2012P000267
Record Dates: First submitted 2013-02-18; First posted 2013-09-23 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — ubiquinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Depending on the patient's ability to swallow pills, patients in the control group will receive a placebo pill or a liquid placebo, which is 50 milliliters of Ensure (a dietary supplement). This will be given every 12 hours for 7 days or until hospital discharge.
  Interventions: Dietary Supplement: Placebo
- Ubiquinol (Experimental): Depending on the patient's ability to swallow pills, patients in the experimental group will receive 200mg of Ubiquinol in either a pill or a liquid. The liquid form of the study med will be mixed with 50 milliliters of Ensure (a dietary supplement) to ensure blinding. This will be given every 12 hours for 7 days or until hospital discharge.
  Interventions: Drug: Ubiquinol

INTERVENTIONS:
Drug: Ubiquinol — Depending on the patient's ability to swallow pills, patients in the experimental group will receive 200mg Ubiquinol in either a pill or a liquid. The liquid form of the study med will be mixed with 50 milliliters of Ensure (a dietary supplement) to ensure blinding. This will be given every 12 hours for 7 days or until hospital discharge.
  Arms: Ubiquinol
Dietary Supplement: Placebo — Depending on the patient's ability to swallow pills, patients in the control group will receive a placebo pill or a liquid placebo, which is 50 milliliters of Ensure (a dietary supplement). This will be given every 12 hours for 7 days or until hospital discharge.
  Other Names: placebo pill or a liquid placebo (Ensure)
  Arms: Control

SUMMARY:
This study aims to determine if Ubiquinol (reduced form of COQ10) will attenuate mitochondrial injury and decrease inflammatory response in patients suffering from sepsis.

DETAILED DESCRIPTION:
Severe sepsis and septic shock are the cause of significant morbidity and mortality worldwide. An estimated 751,000 (3 per 1,000 population) cases of severe sepsis occur in the United States each year, resulting in approximately 215,000 deaths. Septic shock is characterized by hypotension, hypermetabolic state, lactic acidosis, and potentially death. In addition, the economic burden on the health care system for patients suffering from severe sepsis is striking. Weycker et al. report that patients suffering from severe sepsis will require an average of $45,000 dollars of medical care cost on their index admission and up to $78,500 dollars in the first year post-diagnosis. These figures rival such entities as acute myocardial infarction, trauma, and stroke. Whereas a significant amount of research and therapeutic interventions have been focused on the "early hours" of diseases such as acute myocardial infarction, stroke, and trauma, less attention has been given to the initial stages of severe sepsis and septic shock.

Coenzyme Q10 (CoQ10) is a safe and feasible medicinal intervention with a strong scientific rationale for use in septic shock. CoQ10 is a key component of the mitochondria, serving as an electron transport medium between complex I/II and complex III. A lesion at this point in the electron transport chain results in an inadequate production of ATP (adenosine triphosphate) for the cell. In septic shock, CoQ10 levels are profoundly decreased and therefore production of energy may be compromised. CoQ10 has two essential roles in critically ill patients with sepsis: 1) production of ATP and 2) reduction of free oxygen radicals. CoQ10's key role in the electron transport chain may prevent the well-described mitochondrial dysfunction that occurs in patients with septic shock. Thus, these two essential roles form the pathophysiological basis for this proposed study.

In the following proposal, the investigators plan to perform a pilot study to evaluate the capacity for ubiquinol (reduced form of COQ10) to attenuate mitochondrial injury, to attenuate inflammation/vascular endothelial injury, the effect on the human metabolome, and to be absorbed. The overall goal of this line of research will be to determine if CoQ10 will attenuate oxidative injury and improve mitochondrial function leading to overall improved outcome in patients suffering from septic shock. In order to achieve this long-term goal, the investigators propose this pilot and feasibility trial to determine CoQ10 absorption in critical illness, capacity to mitigate inflammatory injury and oxidative injury, and ability to maintain mitochondrial electron transport chain functionality. This pilot study will also provide key feasibility data on blinding and other logistical issues necessary for execution of a larger-scale investigation.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Suspected or confirmed infection
* Presence of 2 or more systemic inflammatory response syndrome (SIRS) criteria
* Admission to the ICU

Exclusion Criteria:

* Under 18 years old
* Current CoQ10 supplementation
* Unable to receive enteral medications
* Would need a nasogastric or orogastric tube solely for the purposes of the study
* Pregnancy, incarceration, mentally disability
* Patient confirmed Comfort measures only, Do not resuscitate (DNR) and/or Do not intubate. Patients with DNR but intubated and being provided full care are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donnino MW, Mortensen SJ, Andersen LW, Chase M, Berg KM, Balkema J, Radhakrishnan J, Gazmuri RJ, Liu X, Cocchi MN. Ubiquinol (reduced Coenzyme Q10) in patients with severe sepsis or septic shock: a randomized, double-blind, placebo-controlled, pilot trial. Crit Care. 2015 Jul 1;19(1):275. doi: 10.1186/s13054-015-0989-3. PMID 26130237

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient was randomized in the placebo group but the blood was accidentally thawed why this patient was excluded. 2 patients were randomized in the Ubiquinol group but never received the treatment (one because of an exclusion criteria and one because of a Boston-wide mass casualty event). These were also excluded.
Period: Overall Study
Arm/Group | Placebo | Ubiquinol
Started | 20 | 21
Completed | 19 | 19
Not Completed | 1 | 2
Not completed — Boston MCI halted research protocol | 0 | 1
Not completed — Discovered an enrollment in other study | 0 | 1
Not completed — Blood samples were accidentally thawed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Patients will receive a placebo pill or a liquid placebo. The liquid placebo is 50 milliliters of Ensure (a dietary supplement). Placebo will be given every 12 hours for 7 days or until hospital discharge.
- Ubiquinol: Patients will receive 200mg of Ubiquinol in either a pill or a liquid. The liquid form of the study med will be mixed with 50 milliliters of Ensure (a dietary supplement) to ensure blinding. This will be given every 12 hours for 7 days or until hospital discharge.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ubiquinol | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64 (14) | 60 (18) | 62 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 8 | 12 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 18 | 33
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 3 | 7
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: CoQ10 Levels
Description: Total CoQ10 levels (mcg/mL) at 24 hours post study drug admission.
Time Frame: 24 hours after study drug administration
Measure: Median (Inter-Quartile Range); unit: (mcg/mL)
Arm/Group | Placebo | Ubiquinol
Number analyzed (Participants) | 19 | 19
(mcg/mL) | 0.38 [0.26 to 0.66] | 0.87 [0.57 to 1.26]

ADVERSE EVENTS:
Time Frame: Hospital stay, average 10 days
Arm/Group | Ubiquinol | Placebo
All-Cause Mortality (participants affected / at risk) | 4/19 | 2/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 1/19 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ubiquinol (N=19) | Placebo (N=19)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No